CLINICAL TRIAL: NCT03869489
Title: Decision Making in Video Games
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Goals changed
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1809016
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Cognitive Change
Keywords: approach motivation; avoidance motivation; transcranial direct current stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Anodal left dorsolateral prefrontal cortex tDCS stimulation (Experimental)
  Interventions: Device: Anodal left dorsolateral prefrontal cortex tDCS stimulation
- Anodal right dorsolateral prefrontal cortex tDCS stimulation (Experimental)
  Interventions: Device: Anodal right dorsolateral prefrontal cortex tDCS stimulation
- Sham tDCS stimulation (Sham Comparator)
  Interventions: Device: Sham tDCS stimulation

INTERVENTIONS:
Device: Anodal left dorsolateral prefrontal cortex tDCS stimulation — Anodal tDCS will be applied to the left dorsolateral prefrontal cortex of participants
  Arms: Anodal left dorsolateral prefrontal cortex tDCS stimulation
Device: Anodal right dorsolateral prefrontal cortex tDCS stimulation — Anodal tDCS will be applied to the right dorsolateral prefrontal cortex of participants
  Arms: Anodal right dorsolateral prefrontal cortex tDCS stimulation
Device: Sham tDCS stimulation — Sham tDCS stimulation will be applied
  Arms: Sham tDCS stimulation

SUMMARY:
The purpose of this study is to determine whether anodal transcranial direct current stimulation (tDCS) applied to the left dorsolateral prefrontal cortex induces approach motivation, and whether anodal tDCS applied to the right dorsolateral prefrontal cortex induces avoidance motivation. This study consists of three experiments: one in which an approach/avoidance video game is validated, one in which the effect of anger and fear on approach/avoidance is studied, and one in which the effect of tDCS is studied. Only the experiment in which the effect of tDCS is studied involves tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing and vision

Exclusion Criteria:

* Left-handedness
* History of seizure, head injury (including neurosurgery), brain injury, diagnosis or a neurological or psychiatric disorder, metal in the head, sensitive scalp
* History of anxiolytic and/or antidepressant medications
* Participation in Experiment #1 or Experiment #2 of the larger study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Avoidance-Approach time difference | 1 year
  Median of the difference between time to approach and time to avoid a stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Applied Brain and Cognitive Sciences, Medford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
N/A. Study withdrawn